CLINICAL TRIAL: NCT05694117
Title: White Box Modeling of Self-Determine Sequence Exercise Program Among Sarcopenic Elderly: Uncovers a Novel Strategy Overcoming Decline of Skeletal Muscle Area
Brief Title: A Study of the Intervention Effect of a Hybrid Exercise Program on Elderly With Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeast Normal University (Other)
Responsible Party: Principal Investigator, Guang Yang, Prof. Dr., Prof.Dr., Northeast Normal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CCEE2019
Record Dates: First submitted 2023-01-11; First posted 2023-01-23 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Sarcopenia
Keywords: sarcopenia; elderly; exercise program; explainable artificial intelligence
MeSH Terms: conditions — Sarcopenia | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- self-determine sequence exercise program (Experimental): The trial was divided into three cycles, and participants were allowed to choose any one of the a Taichi exercise program, a hybrid program of Taichi exercise and resistance training programs, and resistance training as their intervention content before the start of each cycle. Participants who chose Taichi exercise performed one hour of Taichi exercise for each session, while participants who chose a hybrid exercise program of Taichi exercise and resistance training completed Taichi exercise in the first half hour and resistance training for the second half hour. Participants who chose resistance training performed one hour of resistance training. One hour per training session, three times a week for 24 weeks
  Interventions: Behavioral: self-determine sequence exercise program
- resistance training (Experimental): Resistance strength training for resistance exercise and aimed at promoting the greatest hypertrophy response. Training is divided into three cycles, with progressive training load. Resistance exercise intervention three times a week for 24 weeks, one hour each time.
  Interventions: Behavioral: resistance training
- control group (No Intervention): The participants in the control group were introduced by nurses to education about sarcopenia and various methods for preventing it, such as consuming more protein through their diet and participating in greater physical exercise.
- Taichi exercise and resistance training (Experimental): The trial was divided into three cycles, each lasting eight weeks. Participants performed a hybrid program of Taichi exercise and resistance training of varying duration and intensity in each cycle. Each session lasted one hour, three times a week for 24 weeks.
  Interventions: Behavioral: Taichi exercise and resistance training
- Randomly selected exercise program (Experimental): The trial was divided into three cycles, and participants were allowed to choose any one of the a Yijinjing exercise program, a hybrid program of Yijinjing exercise and resistance training programs, and resistance training as their intervention content before the start of each cycle. Participants who chose Yijinjing exercise performed one hour of Yijinjing exercise for each session, while participants who chose a hybrid exercise program of Yijinjing exercise and resistance training completed Yijinjing exercise in the first half hour and resistance training for the second half hour. Participants who chose resistance training performed one hour of resistance training. One hour per training session, three times a week for 24 weeks
  Interventions: Behavioral: Randomly selected exercise program

INTERVENTIONS:
Behavioral: self-determine sequence exercise program — The Taichi exercise utilized the simplified eight styles of Taichi. The resistance training program consisted of three cycles. In the first cycle, investigators used a light load but high repetitions (ranging from 40% to 60% of one repetition maximum and 12-20 repetitions). During the second phase of our training, investigators raised the training load by doing sets of moderate intensity and a medium number of repetitions (ranging from 60% to 80% of one repetition maximum and 5-12 repetitions). In the third cycle, investigators aimed to improve the participants' maximal muscular resistance by using a greater training load and fewer repetitions (ranging from 70% to 85% of one repetition maximum and 5-8 repetitions).
  Arms: self-determine sequence exercise program
Behavioral: resistance training — The resistance training program consisted of three cycles. In the first cycle, investigators used a light load but high repetitions (ranging from 40% to 60% of one repetition maximum and 12-20 repetitions). During the second phase of our training, investigators raised the training load by doing sets of moderate intensity and a medium number of repetitions (ranging from 60% to 80% of one repetition maximum and 5-12 repetitions). In the third cycle, investigators aimed to improve the participants' maximal muscular resistance by using a greater training load and fewer repetitions (ranging from 70% to 85% of one repetition maximum and 5-8 repetitions). Participants in the RTG completed four sets of each movement, with two to three minutes of rest between each set.
  Arms: resistance training
Behavioral: Taichi exercise and resistance training — The training of the Taichi exercise and resistance training group consisted of two cycles, the first cycle was aimed at learning and consolidating Taichi exercise, and the second cycle was aimed at improving and consolidating. The Taichi exercise and resistance training group was scheduled for 30 min of Taichi exercise per training. The resistance training program consisted of three cycles. In the first cycle, investigators used a light load but high repetitions (ranging from 40% to 60% of one repetition maximum and 12-20 repetitions). During the second phase of our training, investigators raised the training load by doing sets of moderate intensity and a medium number of repetitions (ranging from 60% to 80% of one repetition maximum and 5-12 repetitions). In the third cycle, investigators aimed to improve the participants' maximal muscular resistance by using a greater training load and fewer repetitions (ranging from 70% to 85% of one repetition maximum and 5-8 repetitions).
  Arms: Taichi exercise and resistance training
Behavioral: Randomly selected exercise program — Participants in the randomly selected exercise program group who chose Yijinjing exercise were required to complete one hour of Yijinjing exercise training, and those who chose Yijinjing exercise hybrid strength training had to complete half an hour of Yijinjing training. The resistance training program consisted of three cycles. In the first cycle, investigators used a light load but high repetitions (ranging from 40% to 60% of one repetition maximum and 12-20 repetitions). During the second phase of our training, investigators raised the training load by doing sets of moderate intensity and a medium number of repetitions (ranging from 60% to 80% of one repetition maximum and 5-12 repetitions). In the third cycle, investigators aimed to improve the participants' maximal muscular resistance by using a greater training load and fewer repetitions (ranging from 70% to 85% of one repetition maximum and 5-8 repetitions).
  Arms: Randomly selected exercise program

SUMMARY:
Sarcopenia is a geriatric condition characterized by a progressive decrease in skeletal muscle content and loss of muscle function. Resistance exercise, Taichi exercise and the hybrid exercise program consisting of the two aforementioned methods have been demonstrated could increase the skeletal muscle mass of the elderly with sarcopenia. However, note that the above contents may be performed in a different order in a treatment, equally important but less well understood is the sequence in which it should be performed. Surprisingly, the exercise sequence has not been comprehensively investigated. Therefore, investigators designed a self-ordered exercise program combining resistance exercise, tai chi and a hybrid exercise program to investigate whether the decline in skeletal muscle area could be better overcome and the reversal of sarcopenia in elderly with sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

1. satisfied the Asian screening criteria for sarcopenia by the Asian Working Group for Sarcopenia;
2. age higher than 60 but less than 75 years of age.

Exclusion Criteria:

1. with serious illness or breathing failure;
2. with neuro-muscular diseases;
3. taking medication that has an effect on the function of skeletal muscles;
4. with conditions relating to the neurological system or the mental health;
5. in another scheduled training plan.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Using quantitative CT to investigate the change of skeletal muscle area in sarcopenic elderly. | Month 6
  Participants will receive quantitative CT scans before and after the intervention to assess the change from baseline skeletal muscle area at 6 months.
Using a Jamar hydraulic hand dynamometer to investigate change of handgrip in sarcopenic elderly. | Month 6
  Participants will receive a handgrip strength test before and after the intervention to assess the change from baseline handgrip strength at 6 months.
Using a bioelectrical impedance body composition analyzer with a multifrequency device to investigate the change of relative skeletal muscle mass index in sarcopenic elderly. | Month 6
  Participants will receive a relative skeletal muscle mass index test before and after the intervention to assess the change from baseline relative skeletal muscle index at 6 months.

SECONDARY OUTCOMES:
Collect participants' self-evaluation of their life state and physical state. | Month 6
  Participants were asked to write a self-assessment report of no more than 500 words before and after the intervention, including physical status and life status.
Collect video of participants throughout the intervention. | Month 6
  The entire intervention process was videotaped and video of the entire intervention process was collected from the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Guang Yang, Study Chair — Chinese Center of Exercise Epidemiology
Locations (1):
- Chinese Center of Exercise Epidemiology, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wei M, He S, Meng D, Lv Z, Guo H, Yang G, Wang Z. White Box Modeling of Self-Determined Sequence Exercise Program Among Sarcopenic Older Adults: Uncovering a Novel Strategy Overcoming Decline of Skeletal Muscle Area. J Aging Phys Act. 2025 Jun 27:1-13. doi: 10.1123/japa.2024-0123. Online ahead of print. PMID 40581354
- [Derived] He S, Wei M, Meng D, Wang Z, Yang G, Wang Z. Self-determined sequence exercise program for elderly with sarcopenia: A Randomized controlled trial with clinical assistance from explainable artificial intelligence. Arch Gerontol Geriatr. 2024 Apr;119:105317. doi: 10.1016/j.archger.2023.105317. Epub 2023 Dec 21. PMID 38176122